CLINICAL TRIAL: NCT06265064
Title: Can Combination of STOP-Bang Score and Factors Predicting Difficult Intubation Improve Accuracy of Prediction Difficult Mask Ventilation in Obese Patients?
Brief Title: STOP-Bang Score and Factors Predicting Difficult Intubation for Prediction of Difficult Mask Ventilation in Obese Patients
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Petsiri Thaweewan, Principal Investigator, Khon Kaen University
Other Study IDs: KhonKaenUniversity
Record Dates: First submitted 2023-12-10; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Obesity; OSA
Keywords: mask ventilation; general anesthesia
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Difficult mask ventilation: Difficult Mask Ventilation Grading (by Han et al.) Grade 1 mask ventilation can be easily performed by a single person Grade 2 requires the use of equipment such as an oropharyngeal airway Grade 3 necessitates the involvement of two or more personnel for mask ventilation or increasing oxygen flow Grade 4 indicates an inability to perform mask ventilation If the grade is ≥ 3, it signifies difficult mask ventilation
  Interventions: Diagnostic Test: STOP-Bang score >= 3 with factors predicting difficult intubation
- non-difficult mask ventilation: Difficult Mask Ventilation Grading (by Han et al.) Grade 1 mask ventilation can be easily performed by a single person Grade 2 requires the use of equipment such as an oropharyngeal airway Grade 3 necessitates the involvement of two or more personnel for mask ventilation or increasing oxygen flow Grade 4 indicates an inability to perform mask ventilation If the grade is < 3, it signifies non-difficult mask ventilation
  Interventions: Diagnostic Test: STOP-Bang score >= 3 with factors predicting difficult intubation

INTERVENTIONS:
Diagnostic Test: STOP-Bang score >= 3 with factors predicting difficult intubation — patients with STOP-Bang score >= 3 with Mallampati score ≥ 3 or neck circumference >42 cm or mentothyroid distance <6 cm

SUMMARY:
The goal of this prospective observational study is to test combination of STOP-Bang score and factors predicting difficult intubation can improve accuracy of prediction difficult mask ventilation in obese patients that undergoing to elective surgery under general anesthesia.

The main question[s] it aims to answer are:

* Can combination of STOP-Bang score and factors predicting difficult intubation improve accuracy of prediction difficult mask ventilation in obese patients?
* Study about complication after endotracheal tube insertion in obese patients that undergoing to elective surgery under general anesthesia.

Participants who undergoing to elective surgery under general anesthesia will

* Routine preoperative evaluation and ask about STOP bang questions, evaluate neck circumference, Mallampati grade,Thyromental distance (That routine physical examination for anesthetic care pre-operation)
* In operation room, patients will be inducted anesthesia by anesthesiologist (step routine for general anesthesia),observe difficult mask ventilation grading before intubate endotracheal tube and complication after endotracheal tube insertion.

If there is a comparison group:

Researchers will compare obese patients with/without high STOP bang score >=3 point plus factor predicting difficult intubation (Mallampati grade 3-4, Neck circumference > 42 cm, Thyromental distance < 6 cm)to prediction difficult mask ventilation

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25 kg/m2
* Age > 18 years old
* undergoing elective surgery under general anesthesia with endotracheal intubation

Exclusion Criteria:

* History of difficult mask and intubation
* Maxillofacial or upper airway malformation
* History of C-spine disease such as trauma, degeneration
* Pregnancy
* Rapid sequence induction technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Calculation by Diagnotic test that used sensitivity and Specificity of the precedent journal "Accuracy of STOP-Bang Questionnaire in Predicting Difficult Mask Ventilation: An Observational Study by Marium N. Khan , Aliya Ahmed" total population 278 patients
Sampling Method: Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Difficult mask ventilation | After the induction of general anesthesia, observe the assisted mask ventilation. End the collection of the primary outcome before endotracheal tube intubation.
  Difficult Mask Ventilation Grading (by Han et al.) Grade 1 mask ventilation can be easily performed by a single person Grade 2 requires the use of equipment such as an oropharyngeal airway Grade 3 necessitates the involvement of two or more personnel for mask ventilation or increasing oxygen flow Grade 4 indicates an inability to perform mask ventilation If the grade is ≥ 3, it signifies difficult mask ventilation

SECONDARY OUTCOMES:
Resipiratory complication | during mask ventilation until the completion of intubation.
  1. Airway trauma
  2. Desaturation Spo2<90% in 2 minutes
  3. Regurgitation
  4. Aspiration

CONTACTS AND LOCATIONS:
Locations (1):
- KhonKaen University, Nai Muang, Khonkaen, Thailand

IPD SHARING:
Plan to Share IPD: Undecided